CLINICAL TRIAL: NCT05336240
Title: PCOM2 - The Physician Communication Intervention, Version 2.0" for "Linking the Provider Recommendation to Adolescent HPV Vaccine Uptake"
Brief Title: PCOM2 - The Physician Communication Intervention, Version 2.0
Acronym: PCOM2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Kansas Medical Center (Other); San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-4870
Record Dates: First submitted 2022-03-30; First posted 2022-04-20 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: HPV Infection; Preventive Health Services
Keywords: Immunization; Provider Communication; HPV Prevention
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysts on the study team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCOM Standard Arm (Active Comparator): Providers in participating in the PCOM-standard intervention will be trained on optimizing an in-person provider communication technique about HPV vaccination by training primary care providers in a 2-step verbal communication process: 1) to start the HPV vaccine discussion using a "presumptive" format, and 2) to use motivational interviewing (MI) techniques to address parental vaccine hesitancy.
  Interventions: Behavioral: Physician Communication Standard (PCOM-standard)
- PCOM2 Virtual Arm (Experimental): Providers participating in the PCOM2-virtual arm will receive training on this communication method through an adapted virtual model of PCOM-standard.
  PCOM2-Virtual intervention will result in a "shelf ready" intervention and associated "User Manual" that can be easily incorporated into practices broadly to improve the practice's adolescent HPV vaccination rates. PCOM-Virtual arm will then be compared to that of the original PCOM-standard intervention in its efficacy for increasing HPV vaccination among adolescents.
  Interventions: Behavioral: Physician Communication 2 Virtual (PCOM2-virtual)

INTERVENTIONS:
Behavioral: Physician Communication 2 Virtual (PCOM2-virtual) — The PCOM-standard intervention is based off of a provider communication training that utilizes presumptive technique when initiating the vaccine discussion followed by motivational interviewing if a parent continues to show hesitation. While this provider communication technique previously showed success in increasing HPV vaccination uptake, it is neither easy to disseminate nor sustainable due to it's nature of direct, intensive in-person training. Therefore, the intervention is to compare the standard-PCOM intervention to a new, PCOM2 intervention, that will be adapted virtually.
  Arms: PCOM2 Virtual Arm
Behavioral: Physician Communication Standard (PCOM-standard) — The PCOM-standard intervention is based off of a provider communication training that utilizes presumptive technique when initiating the vaccine discussion followed by motivational interviewing if a parent continues to show hesitation. PCOM-standard will be conducted in-person with providers.
  Arms: PCOM Standard Arm

SUMMARY:
Poor quality of primary care providers' vaccine recommendations lead to low adolescent human papillomavirus vaccination rates and hundreds of thousands of adolescents unnecessarily at risk for HPV-associated cancers and diseases. Though a previous provider communication intervention, called PCOM, was found to be effective for increasing adolescent HPV vaccination in primary care, its dissemination is limited by the need for significant research team involvement to teach providers how to use the intervention's components. To address this, investigators propose to develop and test a virtual version of PCOM, use mixed methods to assess contextual factors affecting its use compared to the original PCOM intervention, and develop an optimized version of PCOM for broad dissemination to increase adolescent HPV vaccination nationally.

DETAILED DESCRIPTION:
The overarching goal is to develop a "Virtual" version of the PCOM intervention ("PCOM-Virtual") and compare its efficacy for increasing HPV vaccination among adolescents to that of the original PCOM intervention ("PCOM-Standard"). Using Dissemination & Implementation (D&I) science principles to develop and evaluate the PCOM-Virtual intervention for non-inferiority, investigators anticipate that to have a "shelf ready" intervention and associated "User Manual" that can be easily incorporated into practices broadly to improve the practice's adolescent HPV vaccination rates.

Specific Aims are to: (1) develop the "PCOM-Virtual" intervention using principles of D&I Science; (2) compare the efficacy of "PCOM-Virtual" versus "PCOM-Standard" in improving adolescent HPV vaccine utilization; and (3) examine whether practice, patient and provider characteristics are associated with variability in the efficacy of PCOM-Virtual and PCOM-Standard.

ELIGIBILITY:
Inclusion Criteria:

* Parents: Have an adolescent between the ages of 9-17 years old and receiving adolescent care at an enrolled clinic
* Providers: All providers at participating study practices will be eligible to participate.

Exclusion Criteria:

* Parents: Does not have an adolescent between the ages of 9-17 years old and is not receiving adolescent care at an enrolled clinic
* Providers: Providers who are not at participating study practices

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccination initiation status in 11-12 year olds | Adolescent vaccination initiation status will be assessed among all "active" (seen in the last 12 months) 11 to 12-year-old patients at each practice during the last 12 months of the 24 month intervention period
  The primary outcome to be assessed in the trial is HPV vaccine series initiation among 11-12-year-olds as 11-12 year-olds are the preferred target population for HPV vaccination and the PCOM intervention had its strongest effect on series initiation rather than completion.

SECONDARY OUTCOMES:
HPV series completion among 11-12 year olds | Adolescent vaccination completion status will be assessed among all "active" (seen in the last 12 months) 11 to 12-year-old patients at each practice during the last 12 months of the 24 month intervention period
  Secondary outcome to assess HPV series completion among 11-12-year-olds
HPV vaccination initiation status in 13-17 year olds | Adolescent vaccination initiation status will be assessed among all "active" (seen in the last 12 months) 13-17-year-old patients at each practice during the last 12 months of the 24 month intervention period
  Secondary outcome to assess "catch-up" HPV vaccine series initiation among 13-17-year-olds
HPV series completion among 13-17 year olds | Adolescent vaccination completion status will be assessed among all "active" (seen in the last 12 months) 13-17-year-old patients at each practice during the last 12 months of the 24 month intervention period
  Secondary outcome to assess "catch-up" HPV vaccine series completion among 13-17 year-olds.

CONTACTS AND LOCATIONS:
Overall Officials: Sean O'Leary, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Kansas Medical Center, Wichita, Kansas

IPD SHARING:
Plan to Share IPD: No